CLINICAL TRIAL: NCT05449314
Title: Cultural Adaptation and Validation of Urdu Version of Modified Barthel Index to Assess the Independence of Pakistani Stroke Patients
Brief Title: Reliability and Validity Study of Urdu Version of Modified Barthel Index in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0295
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Stroke
Keywords: Modified Barthel index; Urdu Version; Reliability; Validity; Cerebrovascular Disease; Stroke; Activities of Daily Living
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study is to translate and culturally adapt the modified Barthel index into Urdu language and to investigate the reliability and validity of this scale in Urdu speaking Stroke population for performance evaluation. Also check its correlation with Functional independence measure and Katz index of Activities of Daily Living.

DETAILED DESCRIPTION:
The English version of the Barthel index will be translated and traditionally adapted as prior endorsement. In Activities of Daily Livings disabled stroke population, Urdu Version of Modified Barthel Index will distributed among sixty participants choose by convenience sampling technique based on pre-distinct inclusion and exclusion standards. To test inter and intra-observer reliability of the final Urdu Version of Modified Barthel Index will be completed on the same day, by two observers, and for the inter-observers evaluation, with an interval of 30 minute between the first and the second submission. Third evaluation will be carried out after 7 days by Observer-1, for intra-observer assessment. Data will be entered and analyzed using Statistical Package of Social Sciences Version 24. Core steadiness will be analyzed with Cronbach alpha value. Test-retest reliability will be evaluated using an intra-class correlation coefficient.The Urdu Version of Modified Barthel Index will be evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Male and female both genders
* Adults between the ages of 18 and above
* Patient suffering from Stroke
* Ability to provide informed consent

Exclusion Criteria:

* Suffering from any cardiovascular pathologies
* Any disorder of contagious infections
* Any history of neurological disorders
* Having any spinal deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urdu speaking population with Activities of Daily Living, balance, or gait impairments effected with Stroke
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Modified Barthel Index | 1st day
  Modified Barthel Index explained 10 tasks and scores are according to time and assistance needed by the patient between total score from 0 to 20.Lower score describes greater assistance, and larger score tells less assistance required by patient.
Functional Independence Measure | 1st day
  Functional Independence Measure was developed with 18-items that includes, 7-level ordinal scale, with 1 representing dependence and 7 representing independence. This outcome was designed to measure amount and level of help needed to perform Activities of Daily Living by disabled persons.
Katz index of Activities of Daily Living | 1st day
  The Katz Activities of Daily Living Index assesses basic activities of daily living. It does not assess more advanced activities of daily living. Katz developed another scale for instrumental activities of daily living such as heavy housework, shopping, managing finances and telephoning.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No